CLINICAL TRIAL: NCT01286181
Title: Device-guided Slow Breathing in COPD Patients With Clinically Significant Dyspnea: Phase 2
Brief Title: Device-guided Breathing for Shortness of Breath in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-008433
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: COPD; Dyspnea; Hyperinflation
Keywords: COPD; Biofeedback; Dyspnea; Quality of life; Stress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device-guided slow breathing (Experimental)
  Interventions: Behavioral: Twice daily practice of device-guided slow breathing.

INTERVENTIONS:
Behavioral: Twice daily practice of device-guided slow breathing. — Participants are asked to use the slow-breathing device for 20 minutes twice daily, for 8 weeks. Participants receive weekly telephone calls to monitor device use and are encouraged to use pursed-lips when following the breathing tones of the device while exhaling.

SUMMARY:
Although drug therapies and pulmonary rehabilitation have greatly improved COPD symptoms, as many as 50% of patients with severe COPD have inadequately controlled dyspnea. Device-guided breathing is a behavioral intervention that guides respiratory rates into a therapeutic range; prolongation of the expiratory phase improves hyperinflation, the most significant driver of dyspnea in this population. Device-guided breathing, has no known side-effects, and may represent a cost effective adjunctive treatment for dyspnea in severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Current or former cigarette smokers of at least 10 pack-years
* Clinically significant dyspnea, as determined by a score of at least 2 on the Medical Research Council Dyspnea Score questionnaire (0-4), or through pulmonary function test results of a residual volume (RV) of > 150% predicted or an FEV1 of <65% predicted
* Clinical diagnosis of chronic obstructive pulmonary disease

Exclusion Criteria:

* Unable to use the slow-breathing device due to hearing impairment
* Poor motivation or lack of interest in using the device
* Pulmonary Rehabilitation ordered as a new therapy at the time of enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine effect of increased device-guided breathing on health-related quality of life measures. | 8 weeks
  Pre and post device use measures of dyspnea, health-related quality of life, stress, adn self-efficacy for managing chronic disease will be obtained through self-administered questionnaires.

SECONDARY OUTCOMES:
Evaluate effect of device-guided slow breathing on daily physical activity. | 8 weeks
  Evaluate the effect of a higher intensity of device-guided breathing (20 minutes twice daily for 8 weeks) on daily physical activity, as measured by a gold-standard activity monitor, before and after device use.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States